CLINICAL TRIAL: NCT03220841
Title: Stricture Definition and Treatment (STRIDENT) Drug Therapy Study
Acronym: STRIDENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Australasian Gastro Intestinal Research Foundation (Other); AbbVie (Industry)
Responsible Party: Principal Investigator, Michael Kamm, Professor of Gastroenterology, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StVincentsMelbourneSTRIDENT1
Record Dates: First submitted 2017-07-06; First posted 2017-07-18 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Stricture; Bowel
Keywords: Crohn Disease; Inflammatory Bowel Disease; Intestinal stricture
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Constriction, Pathologic | interventions — Adalimumab; 2-mercaptopurine

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard drug therapy (Active Comparator): Adalimumab monotherapy, Standard Dose induction (160mg at week 0, 80mg week 2 and 40mg fortnightly thereafter)
  Interventions: Drug: Adalimumab Injection; Procedure: Endoscopic balloon dilatation
- Intensive drug therapy (Experimental): Adalimumab in combination with dose optimized thiopurine, Intensive induction (160mg weekly for 4 weeks then 40mg fortnightly). Anti-TNF dose may be increased if ongoing inflammation every 4 months until study endpoint.
  Interventions: Drug: Adalimumab Injection; Drug: Thiopurine; Procedure: Endoscopic balloon dilatation

INTERVENTIONS:
Drug: Adalimumab Injection — Standard dose adalimumab induction and maintenance
Drug: Thiopurine — Dose optimized thiopurine
  Arms: Intensive drug therapy
Procedure: Endoscopic balloon dilatation — Prior to randomization, suitable patients may undergo endoscopic balloon dilatation. Patients undergoing dilatation will be stratified to ensure equal numbers in each study arm.

SUMMARY:
Two thirds of patients with Crohn's disease require intestinal surgery at some time in their life. Intestinal strictures, that is narrowing of the bowel due to inflammation and scarring, are the most common reason for surgery. Despite the high frequency, associated disability, and cost there are no are no treatment strategies that aim to improve the outcome of this disease complication. The STRIDENT (stricture definition and treatment) studies aim to develop such strategies.

DETAILED DESCRIPTION:
Prospective randomised controlled study. Patients with Crohn's Disease who have symptomatic inflammatory intestinal strictures will be randomised to receive standard drug therapy (Anti-TNF monotherapy at standard dose) or intensive drug therapy (Intense Anti-TNF dose induction and escalation for continued inflammation in combination with thiopurine) for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease patients with intestinal stricture(s) identified on CT, MRI or endoscopy.

Exclusion Criteria:

* Acute bowel obstruction requiring urgent surgical intervention
* Deemed by treating physician to have high risk of acute bowel obstruction
* Concurrent active perianal sepsis
* Internal fistulising disease in association with strictures (entero-enteric stulas)
* Low rectal or anal strictures
* Evidence of dysplasia or malignancy from stricture biopsies or adjacent mucosal biopsies
* Patients for whom endoscopy is not suitable due to co-morbidities or clinical state
* Inability to give informed consent
* Suspected perforation of the gastrointestinal tract
* Pregnancy
* Inability to undergo MRI small bowel due to a contraindication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in obstructive symptoms. | 12 months
  Improved pain and or frequency of pain compared to baseline. Obstructive symptoms determined by prospective diary documenting number of episodes of pain in previous 2 weeks and severity of the pain episodes using four-level Likert scale.

SECONDARY OUTCOMES:
Improvement in symptoms | 4, 8 and 12 months
  Improved pain and or frequency of pain compared to baseline. Obstructive symptoms determined by prospective diary documenting number of episodes of pain in previous 2 weeks and severity of the pain episodes using four-level Likert scale.
Improvement in biochemical inflammatory parameters | 12 months
  Serum CRP and fecal calprotectin
Improvement in imaging parameters (Intestinal ultrasound) | 12 months
  Limberg's score
Improvement in imaging parameters | 12 months
  Modified MaRIA score
Surgery | 12 months
  The number of patients that require surgical resection of stricture due to failure of drug therapy.
Improvement in patient reported outcomes (PROs) | 12 months
  SF36
Improvement in patient reported outcomes (PROs) | 12 months
  IBDQ

OTHER OUTCOMES:
Treatment Failure | 12 months
  Number of patients who drop out of the study because of clinical symptoms, acute bowel obstruction, unscheduled endoscopic or surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wright, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne; Bronte Holt, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne; Michael Kamm, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St. Vincent's Hospital Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovett GC, Schulberg JD, Hamilton AL, Wright EK, Holt BA, Sutherland TR, Ross AL, Kamm MA. Long-term Results of Drug Treatment for Crohn's Disease Strictures. Clin Gastroenterol Hepatol. 2025 Sep 17:S1542-3565(25)00805-5. doi: 10.1016/j.cgh.2025.09.014. Online ahead of print. PMID 40972879
- [Derived] Lovett GC, Schulberg JD, Hamilton AL, Wright EK, Sutherland TR, Ross AL, Kamm MA. Crohn's Disease Stricture Response to Treatment Assessed with Magnetic Resonance Imaging and Intestinal Ultrasound: STRIDENT Randomized Trial. Inflamm Bowel Dis. 2025 Oct 1;31(10):2777-2786. doi: 10.1093/ibd/izaf073. PMID 40339148
- [Derived] Schulberg JD, Wright EK, Holt BA, Hamilton AL, Sutherland TR, Ross AL, Vogrin S, Miller AM, Connell WC, Lust M, Ding NS, Moore GT, Bell SJ, Shelton E, Christensen B, De Cruz P, Rong YJ, Kamm MA. Intensive drug therapy versus standard drug therapy for symptomatic intestinal Crohn's disease strictures (STRIDENT): an open-label, single-centre, randomised controlled trial. Lancet Gastroenterol Hepatol. 2022 Apr;7(4):318-331. doi: 10.1016/S2468-1253(21)00393-9. Epub 2021 Dec 8. PMID 34890567